CLINICAL TRIAL: NCT00081276
Title: A Phase II Evaluation Of Triapine (NCI-Supplied Agent: NSC #663249, IND #68338) In Combination With Cisplatin (Commercially Available: NSC # 119875) In The Treatment Of Recurrent Or Persistent Platinum-Resistant Ovarian Or Primary Peritoneal Carcinoma
Brief Title: 3-AP and Cisplatin in Treating Patients With Recurrent or Persistent Platinum-Resistant Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02585; GOG-0126O; U10CA027469 (NIH); CDR0000360854 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; Cisplatin

ARMS (1):
- Treatment (triapine and cisplatin) (Experimental): Patients receive 3-AP IV over 2 hours on days 1-4 and cisplatin IV over 1 hour on days 2 and 3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: triapine; Drug: cisplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as 3-AP and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. This phase II trial is studying how well giving 3-AP together with cisplatin works in treating patients with recurrent or persistent platinum-resistant ovarian epithelial cancer or primary peritoneal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of 3-AP and cisplatin in patients with recurrent or persistent platinum-resistant ovarian epithelial or primary peritoneal cancer.

II. Determine the toxicity of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine the duration of progression-free survival and overall survival in patients treated with this regimen.

II. Determine the effects of prognostic variables, including initial performance status, age, and mucinous (or clear cell) histology, in these patients.

OUTLINE: This is a non-randomized study.

Patients receive 3-AP IV over 2 hours on days 1-4 and cisplatin IV over 1 hour on days 2 and 3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for 5 years.

PROJECTED ACCRUAL: A total of 23-48 patients will be accrued for this study within 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial or primary peritoneal cancer

  * Recurrent or persistent disease
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Outside a previously irradiated field
* Received 1 prior platinum-based chemotherapy regimen (e.g., carboplatin, cisplatin, or other organoplatinum compound) for primary disease

  * Initial treatment may have included high-dose, consolidation, or extended therapy after surgical or non-surgical assessment
* Considered platinum resistant or refractory, according to 1 of the following criteria:

  * Treatment-free interval of less than 6 months after platinum-based therapy
  * Disease progression during platinum-based therapy
* Ineligible for any higher priority GOG protocol
* Performance status - GOG 0-2 (for patients who received 1 prior treatment regimen)
* Performance status - GOG 0-1 (for patients who received 2 prior treatment regimens)
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No serious cardiac disease
* No prior myocardial infarction
* No uncontrolled congestive heart failure
* No pulmonary disease requiring oxygen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Neuropathy (sensory and motor) ≤ grade 1
* No active infections requiring antibiotics
* No hearing impairment
* No known G6PD deficiency
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* At least 3 weeks since prior biologic or immunologic agents for malignant tumor
* One prior non-cytotoxic regimen (e.g., monoclonal antibodies, cytokines, or small-molecule inhibitors of signal transduction) allowed
* See Disease Characteristics
* One prior paclitaxel-containing regimen allowed
* No prior 3-AP
* No other prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimens
* Recovered from prior chemotherapy
* At least 1 week since prior hormonal therapy for malignant tumor
* Concurrent hormone replacement therapy allowed
* No prior radiotherapy to more than 25% of marrow-bearing areas
* Recovered from prior radiotherapy
* Recovered from prior surgery
* No prior cancer therapy that contraindicates receiving study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-07; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Frequency and duration of objective response assessed using RECIST criteria | Up to 5 years
Frequency and severity of observed adverse effects assessed using CTCAE version 3.0 | Up to 5 years

SECONDARY OUTCOMES:
Duration of progression-free survival | From study entry until disease recurrence, death or date of last contact, assessed up to 5 years
Duration of overall survival | From study entry to death or date of last contact, assessed up to 5 years
Prognostic variables (e.g., initial performance status, age, and mucinous [or clear cell] histology) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Usha, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kunos C, Radivoyevitch T, Abdul-Karim FW, Fanning J, Abulafia O, Bonebrake AJ, Usha L. Ribonucleotide reductase inhibition restores platinum-sensitivity in platinum-resistant ovarian cancer: a Gynecologic Oncology Group Study. J Transl Med. 2012 Apr 27;10:79. doi: 10.1186/1479-5876-10-79. PMID 22541066